CLINICAL TRIAL: NCT01791673
Title: Efficacy and Safety of Circular Cyclocoagulation Using High Intensity Focused Ultrasound With EYEOP1 Device in Glaucoma Patients. Prospective Multicenter Clinical Trial.
Brief Title: Circular Cyclocoagulation Using HIFU With EYEOP1 Device in Glaucoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EyeTechCare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EYEMUST-3
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2013-02

CONDITIONS: Glaucoma
Keywords: Glaucoma; Cyclocoagulation; HIFU - High Intensity Focused Ultrasound; Ciliary Body
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound Glaucoma treatment (Experimental): Cyclocoagulation using High Intensity Focused Ultrasound (HIFU)
  Interventions: Device: Ultrasound glaucoma treatment

INTERVENTIONS:
Device: Ultrasound glaucoma treatment — Ultrasound glaucoma treatment with EYEOP1 device
  Other Names: UCP

SUMMARY:
The aim of the study is to evaluate the effectiveness and the safety of the cyclocoagulation using HIFU in glaucoma patients

ELIGIBILITY:
Inclusion Criteria:

* Primary Open-angle glaucoma included pseudo-exfoliative glaucoma and pigmentary glaucoma
* IOP > 21 mm Hg on glaucoma medications, and indicated for filtering glaucoma surgery
* Patient must be aged 18 years and more
* No previous cyclophotocoagulation procedure in the eye
* No previous laser treatment in the eye during the 3 months before HIFU procedure

Exclusion Criteria:

* History of previous glaucoma surgery with implantation of glaucoma drainage device in the study eye
* History of ocular or retrobulbar tumor
* retinal detachment, choroidal hemorrhage or detachment
* Ocular infectious diseasee within 14 days before HIFU procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Success rate : Proportion of eyes that achieve an IOP of > 5 mmHg and <21 mmHg or an IOP reduction > 20% | up to 12 months
  Success rate = complete success rate (achieved without ocular hypotensive medication) + qualified success (achieved with ocular hypotensive medication)

SECONDARY OUTCOMES:
Average change in IOP (mm Hg) | 3, 6 and 12 months
Percentage change in IOP from baseline | 3, 6 and 12 months
Average change in glaucoma hypotensive medications | 3, 6 and 12 months
Incidence of device and procedure-related complications during follow-up | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe DENIS, MD, Principal Investigator — Croix Rousse University Hospital
Locations (5):
- France (5):
  - University Hospital, Dijon
  - Michallon University Hospital, Grenoble
  - Huriez University Hospital, Lille
  - Croix Rousse University Hospital, Lyon
  - HIA - Val de Grace Hospital, Paris